CLINICAL TRIAL: NCT03876002
Title: Evaluation of Microglial Activation Using the PET Imaging Ligand [18F]PBR06 in Patients With Amyotrophic Lateral Sclerosis Compared to Healthy Volunteers
Brief Title: Evaluation of Microglial Activation in ALS With [18F]PBR06 (Peripheral Benzodiazepine Receptor-06) PET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Molecular NeuroImaging (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: [18F]PBR06
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Healthy Volunteers; Amyotrophic Lateral Sclerosis
Keywords: HV; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — N-fluoroacetyl-N-(2,5-dimethoxybenzyl)-2-phenoxyaniline

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]PBR06 (Experimental): To perform kinetic modeling using plasma-based (metabolite corrected plasma concentration) or reference region based methods or simplified quantification methods to assess the ability of [18F]PBR06 PET to measure microglial activation in brain.
  Interventions: Drug: [18F]PBR06

INTERVENTIONS:
Drug: [18F]PBR06 — Subjects will undergo PET imaging using 1 single intravenous (IV) injection of [18F]PBR06, a PET radioligand for evaluation of microglial activation in the brain. PBR06 will be injected intravenously as a bolus at a dose of no more than 5.5mCi (millicurie).

SUMMARY:
The overall goal of this protocol is to evaluate microglial activation in the brain using [18F]PBR06 in patients with amyotrophic lateral sclerosis (ALS).

DETAILED DESCRIPTION:
The overall goal of this protocol is to evaluate microglial activation in the brain using [18F]PBR06 in patients with amyotrophic lateral sclerosis (ALS). The specific objectives are:

* To measure the dynamic uptake and washout of [18F]PBR06 (Peripheral benzodiazepine receptor-06) in brain using positron emission tomography (PET) in patients with ALS and healthy volunteers (HV).
* To evaluate test/retest reliability of the tracer binding parameters in patients with ALS and HV.
* To evaluate the correlation of [18F]PBR06 binding with ALS disease clinical severity (ALSFRS-R, upper motor neuron burden (UMNB) and Ashworth Score), clinical disease sub-categorization, and other clinical data.
* To perform kinetic modeling using plasma-based (metabolite corrected plasma concentration) or reference region based methods or simplified quantification methods to assess the ability of [18F]PBR06 PET to measure microglial activation in brain.
* To acquire safety data following injection of [18F]PBR06.

ELIGIBILITY:
Inclusion Criteria (for all subjects):

* Written informed consent must be obtained before any assessment is performed.
* Provide signed and dated written informed consent.
* Female subjects must be documented by medical records or physician's note to be either surgically sterile (by means of hysterectomy, bilateral oophorectomy, or tubal ligation) or post-menopausal for at least 1 year or, if they are of child-bearing potential, must commit to the use of a barrier method of contraception for the study duration,
* Male subjects and their partners of childbearing potential must commit to the use of a barrier method of contraception for the study duration.
* Male subjects must not donate sperm for the study duration.
* Able to lie supine on camera bed for a reasonable period of time.
* Willing and able to cooperate with study procedures.
* Women of child bearing potential must have a negative pregnancy test at screening.

Inclusion criteria specific to healthy volunteer subjects:

* Males and females aged 45-80 years, healthy with no clinically relevant finding on physical examination at screening and upon reporting for the [18F]PBR06 imaging sessions.
* No family history of ALS or frontotemporal dementia.
* C-reactive protein level ≤10 mg/dL Inclusion criteria specific to ALS subjects
* Males and females aged 18 to 80 years.
* Sporadic or familial ALS diagnosed as possible, laboratory-supported probable, probable, or definite as defined by the modified El Escorial criteria;
* Subjects with a diagnosis of possible ALS must have upper motor neuron (UMN) signs to be eligible
* ALS cognitive behavioral screen score >10 on the cognitive scale and/or >32 on the behavioral scale;
* Forced vital capacity of ≥40%; or if in the opinion of the investigator can lay flat for up to 90 minutes. If an forced vital capacity (FVC) has been performed within the past 6 months; this data may be used at the discretion of the investigator.
* Medications for ALS subjects should be stable for 30 days prior to the Screening Visit and remain unchanged during the subject's participation in the study.

Exclusion Criteria (for all subjects):

* Low affinity translocator protein (TSPO) binders determined by having a Thr/Thr polymorphism in the TSPO gene at screening.
* Treatment with immunosuppressive agents (eg. prednisone, solumedrol) within 30 days of baseline and follow-up imaging.Treatment with anti-inflammatory agents including any medications in the following classes of NSAIDS: carboxylic acids, enolic acids, cyclooxygenase (COX) II Inhibitors within 14 days of baseline and follow-up imaging. Treatment with benzodiazepines within 5 half-lives prior to any [18F]PBR06 imaging visit.
* For subjects undergoing arterial line placement, treatment with any antihemostasis medication (e.g., warfarin, heparin, thrombin inhibitors, Factor Xa inhibitors, streptokinase, urokinase, tissue plasminogen activators) within 2 weeks of the planned arterial line placement of either the baseline or follow-up imaging.
* For subjects undergoing arterial line placement, a Modified Allen's test indicating insufficient ulnar artery blood supply to the hand.
* Current or prior history of alcohol or drug abuse.
* Current tobacco use including cigarettes, cigars, and chewing tobacco, or nicotine-containing products such as gum, patch, or "electronic cigarettes".
* Positive urine drug screen or urine cotinine screen, with the exception of tetrahydrocannabinol (THC) in ALS subjects for whom medical marijuana is prescribed.
* Laboratory tests with clinically significant abnormalities and/or clinically significant unstable medical illness.
* Subject has received an investigational therapeutic within 30 days prior to screening.
* Radiation exposure over the past year (including prior participation in other research protocols, clinical care or participation in this study) exceeding the effective dose of 50 millisievert (mSv), which would be above the acceptable annual limit established by the US Federal Guidelines.
* Pregnancy, lactating or breastfeeding.
* Evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Unsuitable veins for repeated venipuncture.
* MRI exclusion criteria include: Findings that may interfere with interpretation of the [18F]PBR06 PET imaging, including but not limited to: significant cortical cerebrovascular disease, infectious disease, space-occupying lesions, hydrocephalus or other abnormalities associated with central nervous system (CNS) disease.
* Contraindications to MRI imaging, including but not limited to: Implants such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, CNS aneurysm clips and other medical implants that have not been certified for MRI, or history of claustrophobia, which in the opinion of the investigator is severe and prohibits imaging.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-06-28 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

PRIMARY OUTCOMES:
Time-activity data | 1 year
  Time-activity data will be analyzed with 2-tissue compartment model, using the radiometabolite-corrected plasma input function. To correct the brain data for its vascular component, radioactivity in serial whole blood will be measured and then subtracted from the PET measurements. Non-invasive simple tissue ratio methods will also be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: David Russell, M.D., Ph. D, Principal Investigator — Molecular NeuroImaging
Locations (1):
- Molecular NeuroImaging, LLC, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
individual patient data (IPD) that underlie results in any publication will be made accessible for other researchers. All text, tables, figures and appendices will be deidentified. Other documents that will be available include the study protocol, statistical analysis plan, and analytic codes. The data will become available beginning 3 months and ending 5 years article publication via a third-party website (link will be provided). Researchers who provide a methodological sound proposal and aims for intended use of the data will be granted access and will be required to sign a data access agreement. Proposals should be directed to the Study Principal Investigator David Russell, M.D. Ph.D., at david.russell@invicro.com.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available beginning 3 months and ending 5 years article publication.
Access Criteria: Researchers who provide a methodological sound proposal and aims for intended use of the data will be granted access and will be required to sign a data access agreement. Proposals should be directed to the Study Principal Investigator David Russell, M.D. Ph.D., at david.russell@invicro.com.